CLINICAL TRIAL: NCT05856292
Title: Improving Cancer Pain Management Through Teach-Back Educational Approach for Patients and Primary Caregivers: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarumanagara University (Other)
Responsible Party: Principal Investigator, Ricky Dosan, Principal Investigator, Tarumanagara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TarumanagaraU
Record Dates: First submitted 2023-04-11; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Cancer Pain
Keywords: Cancer Pain; Education
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Intervention Model Description: Group 1: Placebo Group 2: Teach-Back
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach-Back (Experimental): The intervention group were educated using the standard educational method with the addition of Teach-back enhancement. It consists of 5 steps: Triage, Tools, Take Responsibility, Tell Me, and Try Again. The Triage, Tools, and Try Again focus on effective information delivery, while the Take Responsibility and Tell Me evaluate the patient's ability to receive the information
  Interventions: Other: Teach Back
- Non-Teach-Back (Placebo Comparator): No educational intervention, just standard educational methods
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Teach Back — Standard cancer pain educational intervention enhanced with teach-back method
  Arms: Teach-Back
Other: Placebo — Standard cancer pain educational intervention without enhancement
  Arms: Non-Teach-Back

SUMMARY:
This randomized prospective quantitative pilot study compared teach-back method to standardized educational method in patient and caregiver to improve cancer pain management

DETAILED DESCRIPTION:
Even though there are comprehensive guidelines for cancer pain management, pain control among cancer patients and survivors is often suboptimal due to undertreatment. According to recent studies, the addition of educational interventions could improve pain relief in cancer patients. Both patients and family caregivers play an important role in delivering cancer pain self-management, especially at home. Providing knowledge for cancer pain management with optimal intervention could improve patient and caregiver outcomes.

The Teach-back method, where patients and family caregivers are asked to repeat the instruction they've received from their health care professionals, can assess patients' understanding, repeat or modify the educational material if comprehension is not demonstrated. This pilot study compared the addition of the Teach-back method for cancer patients and their caregivers and its relation to cancer pain management.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe pain (pain scale 4 and above)
* ≥18 years old
* Signed the informed consent
* Willing to cooperate until the end of studies
* The patient is fully conscious and able to communicate well
* Cared by a family caregiver
* Family caregiver able to fully function as a caregiver

Exclusion Criteria:

* Near-death (dying) stage
* Not willing to cooperate until the end of studies
* Altered mental status and communication difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Cancer pain management | one month
  Quality of cancer pain management. Patient Global Impression Change (PGIC) scale is used to measure the overall quality of life and satisfaction as a conclusion toward the intervention

SECONDARY OUTCOMES:
Health Literacy | one month
  using Health Literacy Short Form Survey Questionnaire (HLS-EU-SQ10-IDN) to measure the change in health literacy
Pain Level | weekly up to one month
  using Brief Pain Inventory (BPI) to measure the change in pain level
Distress | weekly up to one month
  using distress thermometer to measure change in distress
Belief | one month
  using Barriers Questionnaire (BQ-13) to measure change in belief

CONTACTS AND LOCATIONS:
Locations (1):
- Dharmais National Cancer Centre, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No